CLINICAL TRIAL: NCT06968858
Title: First-in-human Study to Assess the Clinical Feasibility, Safety, and Performance of the α Prototype of the NIMBLE System for Diagnosing Complications in Intracoronary Stents. NIMBLE-I Study.
Brief Title: Pilot Study of the α Prototype NIMBLE System: Feasibility, Safety, and Initial Performance in Non-Invasive Detection of Coronary In-Stent Restenosis
Acronym: NIMBLE-I
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Nimble Diagnostics S.L. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: NDX-0001
Record Dates: First submitted 2025-04-24; First posted 2025-05-13 (Actual); Last update posted 2025-05-13 (Actual); Status verified 2025-05

CONDITIONS: In-stent Restenosis; Stent Fracture; Stent Complication
Keywords: non-invasive; microwave; prototype; nimble; in-stent restenosis

STUDY DESIGN:
Intervention Model Description: All enrolled participants will undergo a single, non-invasive measurement with the NIMBLE System prior to their scheduled invasive coronary angiography. No randomization or comparison groups are included. A subset of 30 participants will also undergo optical coherence tomography (OCT) to provide additional reference data. Usability and safety assessments will be conducted based on operator and patient feedback.
Masking Description: The NIMBLE System measurement is performed prior to the invasive coronary angiography, ensuring that the operator conducting the NIMBLE assessment is blinded to the results of the reference standard (angiography and, when applicable, OCT). This approach minimizes potential diagnostic bias and preserves the objectivity of the non-invasive measurement.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental (Experimental): Patients undergoing NIMBLE System measurement prior to coronary angiography
  Interventions: Diagnostic Test: NIMBLE test

INTERVENTIONS:
Diagnostic Test: NIMBLE test — Non-invasive assessment of ISR with the NIMBLE System (Microwave Interferometry)

SUMMARY:
The NIMBLE-I study is a prospective, unicentric, single arm, feasibility clinical trial designed to evaluate a novel medical device for the non-invasive monitoring of coronary stents. The study is being conducted at the Hospital Germans Trias i Pujol in Badalona, Spain, under the supervision of Dr. Oriol Rodríguez Leor, an experienced interventional cardiologist. It is sponsored by NIMBLE Diagnostics, a company developing the NIMBLE system-a non-ionizing, non-invasive prototype based on microwave interferometry (MWI).

The motivation behind the study stems from the clinical challenge of detecting in-stent restenosis (ISR), a common complication following stent implantation that affects up to 10% of patients. Current diagnostic methods typically rely on invasive procedures such as coronary angiography or intravascular imaging, which are resource-intensive and carry procedural risks. The NIMBLE system has the potential to address this need by providing a safe, fast, and non-invasive alternative capable of detecting structural changes around coronary stents.

The primary objective of the NIMBLE-I study is to assess the technical feasibility of the NIMBLE device in a real-world clinical setting. Secondary objectives include evaluating the safety of the device, generating preliminary data on its effectiveness by comparing its measurements with those obtained from invasive coronary angiography-the reference standard for diagnosing ISR-and collecting usability data to inform improvements in future versions of the device.

The study is designed to enroll up to 120 patients of whom 30 will undergo an OCT examination to evaluate the ability of the α prototype to measure ISR. Participants must be adults with previously implanted coronary stents who present with symptoms suggestive of ISR-such as chest pain or ischemic changes on an electrocardiogram-and are already scheduled for diagnostic angiography. Patients with contraindications such as pregnancy, implanted electronic devices (like pacemakers), or anatomical limitations that preclude correct device positioning will be excluded.

The procedure begins with obtaining informed consent from eligible patients. Prior to the scheduled angiographic procedure, the NIMBLE system is used to perform a non-invasive scan. The device, which includes biocompatible transducers, is placed externally over the patient's chest at the level of the coronary stent. Data acquisition does not interfere with standard clinical care. After the NIMBLE scan, patients proceed with their routine coronary angiography as per standard of care. Importantly, operators performing the angiography remain blinded to the results of the NIMBLE device.

Data analysis will focus on two main areas. The primary endpoint is the successful completion of NIMBLE measurements without device-related adverse events. Secondary endpoints include the agreement between NIMBLE output-specifically, a calculated metric called %RIS (percent restenosis intrastent)-and angiographic findings. Statistical methods will be applied to assess sensitivity, specificity, correlation, and agreement between modalities. Usability feedback from clinical operators will also be collected to inform future device iterations.

The study complies with all applicable regulatory and ethical guidelines, including ISO 14155 and the European Medical Device Regulation (MDR 2017/745). It has been approved by the relevant ethics committee and competent authority before its launch. Each patient's data will be anonymized and handled according to Good Clinical Practice (GCP) standards.

Expected outcomes from the NIMBLE-I study include confirmation that the device can be safely and effectively used in a clinical context and that its diagnostic output correlates with invasive imaging findings. Positive results will lay the groundwork for a pivotal clinical trial and advance the development of a tool that could significantly improve the follow-up of patients with coronary stents. Ultimately, this technology could reduce the need for invasive procedures and enable earlier detection of stent-related complications in an outpatient setting.

DETAILED DESCRIPTION:
The NIMBLE-I study is a prospective, single-center, single-arm pilot clinical trial designed to assess the feasibility, safety, usability, and preliminary diagnostic performance of the NIMBLE prototype system. This study represents a significant step forward in the development of non-invasive tools for the detection of complications associated with coronary stents. It is sponsored by NIMBLE Diagnostics and takes place at the Hospital Germans Trias i Pujol in Badalona, Spain, under the leadership of Dr. Oriol Rodríguez Leor, an expert in interventional cardiology.

The rationale behind this study lies in the persistent clinical challenge of in-stent restenosis (ISR)-the re-narrowing of a coronary artery segment within a previously implanted stent. ISR continues to affect 5-10% of all percutaneous coronary intervention (PCI) cases despite advances in stent design and pharmacological therapy. Typically, ISR is diagnosed through invasive procedures such as coronary angiography or intravascular imaging (e.g., IVUS or OCT), which involve patient risk, high cost, and hospital-based infrastructure. The NIMBLE system, which employs microwave interferometry (MWI), offers a novel, non-invasive, and non-ionizing approach aimed at detecting tissue-level changes and structural anomalies suggestive of ISR. The system functions through external thoracic placement of signal transducers, which detect signal interactions with implanted metallic stents.

The primary objective of the NIMBLE-I trial is to demonstrate the technical feasibility and safety of using the NIMBLE prototype in real clinical settings. A secondary objective is to explore the potential of the device in identifying patients with significant ISR by comparing its diagnostic outputs with those of conventional invasive coronary angiography, the current standrd of care. Also, the study will alow to identify potential areas for improvement of the device.

The study plans to include up to 120 patients, of whom 30 will undergo an OCT examination to evaluate the ability of the α prototype to measure ISR. All participants must be adults with a previously implanted coronary stent and present with clinical symptoms suggestive of stent-related complications, such as chest pain or ischemic changes on an ECG. Only patients already scheduled to undergo a diagnostic coronary angiogram as part of their routine care will be eligible. Key exclusion criteria include pregnancy, the presence of implanted electronic medical devices that could interfere with microwave signals (such as pacemakers or defibrillators), or any anatomical constraints that would make transducer placement ineffective.

The clinical procedure begins with the acquisition of written informed consent. Prior to undergoing coronary angiography, each patient is evaluated with the NIMBLE device. The transducers are positioned externally on the patient's chest, over the region of the implanted stent. The measurement session is brief and completely non-invasive, with no interference in the patient's scheduled care. The system captures signal patterns and calculates a parameter which reflects potential stent obstruction. Once the NIMBLE scan is complete, the patient proceeds to undergo standard invasive angiography. Importantly, the interventional team conducting the angiography is blinded to the NIMBLE results to maintain the objectivity of comparative data.

The study's primary endpoint is the successful acquisition of data using the NIMBLE system and without the occurrence of any adverse event. The secondary endpoints include the comparison of RIS values with angiographic findings, the determination of diagnostic performance metrics such as sensitivity and specificity, and the collection of usability data from clinicians interacting with the device. The evaluation will include both descriptive and comparative statistics, and an interim analysis may be conducted following the initial patient roll-in phase.

The NIMBLE-I study follows all relevant ethical and regulatory standards, including the principles of the Declaration of Helsinki, ISO 14155 for clinical investigation of medical devices, and the EU Medical Device Regulation (MDR 2017/745). All procedures have been reviewed and approved by the local ethics committee and competent health authority. Patient confidentiality and data protection are ensured in accordance with Good Clinical Practice (GCP) guidelines.

The anticipated outcome of this study is the validation of the NIMBLE prototype as a safe and technically reliable tool that can be integrated into the clinical workflow for evaluating coronary stents. A successful pilot study will not only support the technical claims of the system but also provide essential data for the design of a larger pivotal clinical trial. Ultimately, the NIMBLE system could transform the monitoring paradigm of coronary stents by allowing non-invasive, outpatient follow-up, potentially reducing healthcare costs and procedural risks while improving patient comfort and diagnostic accuracy.

ELIGIBILITY:
Inclusion Criteria:

* Prior implantation of one or more coronary stents
* Clinical symptoms suggestive of stent failure (e.g., chest pain, ischemic ECG changes)
* Undergoing scheduled coronary angiography
* Informed consent provided

Exclusion Criteria:

* Pregnancy
* Implanted electronic devices (e.g., pacemakers) that may interfere with MWI
* Inability to provide consent
* Chest conditions preventing correct positioning of the device

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-09-12 (Actual); Primary Completion 2025-09 (Estimated); Study Completion 2025-10 (Estimated)

PRIMARY OUTCOMES:
Feasibility | prior angiography
  Feasibility will be assessed by the proportion of enrolled patients in whom the NIMBLE System measurement can be successfully completed and a usable diagnostic output is obtained.
Safety | 7 days after Nimble test
  Absence of device-related adverse events

SECONDARY OUTCOMES:
Performance | DWithin 24 hours before invasive coronary angiography (single time point assessment)
  The performance of the α prototype of the NIMBLE System will be evaluated by comparing its diagnostic measurements to those obtained through invasive coronary angiography, which is considered the clinical reference standard for identifying ISR.
Usability | User (operator) questionnaire will be administered immediately after the NIMBLE System measurement in the first and last enrolled patients. Patient questionnaire will be administered to every participant immediately after their NIMBLE measurement, on the
  Usability will be assessed through a structured questionnaire completed by the clinical operator. Additional qualitative feedback from operators may also be collected to evaluate ease of use, setup time, and integration into the clinical workflow. The patient usability component is also evaluated through a brief post-procedure questionnaire assessing perceived comfort, clarity of instructions, and overall acceptability of the NIMBLE System.

CONTACTS AND LOCATIONS:
Overall Officials: Oriol Rodriguez-Leor, MD, PhD, Principal Investigator — Germans Trias i Pujol Hospital
Locations (1):
- Hospital Universitari Germans Trias i Pujol, Badalona, Catalonia, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: NIMBLE Diagnostics webpage — https://www.dxnimble.com/